CLINICAL TRIAL: NCT01420861
Title: Open Label Study of the Effect of GTx-758 on Serum PSA and Free Testosterone Levels in Men With Castration Resistant Prostate Cancer and Maintained on Androgen Deprivation Therapy
Brief Title: GTx-758 on Serum Prostate-specific Antigen (PSA) in Men With Castrate Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Clinical Hold
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: G200707
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: castrate resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-fluoro-N-(4-fluorophenyl)-4-hydroxy-N-(4-hydroxyphenyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1000 mg GTx-758 BID (Experimental): subjects will receive daily doses of 1000 mg GTx-758
  Interventions: Drug: GTx-758

INTERVENTIONS:
Drug: GTx-758 — two GTx 758 tablets per day

SUMMARY:
The purpose of this study is to assess the effect of GTx-758 on Serum Prostate-specific antigen (PSA) levels in men with castrate resistant prostate cancer who are maintained on androgen deprivation therapy (Serum PSA response and Serum PSA progression)

ELIGIBILITY:
Inclusion Criteria:

1. Be over 18 years of age
2. Be able to communicate effectively with the study personnel
3. Have histologically confirmed prostate cancer
4. ECOG performance status of 0 to 2
5. Have been treated with ADT(chemical or surgical) for at least 6 months
6. Have castrate level of serum total testosterone (<50 ng/dL)
7. Have a history of serum PSA response after initiation of ADT, serum PSA response is at least a 90% reduction in serum PSA to <10 ng/mL OR undetectable level of serum PSA (less tan or =0.2 ng/mL)
8. Have rising serum PSA on two successive assessments at least 2 weeks apart and serum PSA levels ≥ 2 ng/mL or 2ng/mL and a 25% increase over the nadir after the initiation of ADT
9. Be continued on androgen deprivation therapy throughout this study
10. Give written informed consent prior to any study specific procedures
11. Subjects must agree to use acceptable methods of contraception:

oIf their female partners are pregnant or lactating acceptable methods of contraception from the time of the first administration of study medication until 3 months following administration of the last dose of study medication must be used. Acceptable methods are: Condom used with spermicidal foam/gel/film/cream/suppository. If the subject has undergone surgical sterilization (vasectomy with documentation of azospermia) a condom with spermicidal foam/gel/film/cream/suppository should be used. oIf the male subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 3 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e. barrier method of contraception], surgical sterilization (vasectomy with documentation of azospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}. oIf the female partner has undergone documented tubal ligation (female sterilization), a barrier method {condom used with spermicidal foam/gel/film/cream/suppository} should also be used. oIf the female partner has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS) and a barrier method {condom with spermicidal foam/gel/film/cream/suppository} should also be used.

Exclusion Criteria:

1. Known hypersensitivity or allergy to estrogen or estrogen like drugs;
2. Have symptomatic metastatic prostate cancer
3. Any disease or condition (medical or surgical) which might compromise the hematologic, cardiovascular, endocrine, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk;
4. History of abnormal blood clotting, Factor V Leiden clotting disorder, thrombotic disease (venous or arterial thrombotic events such as history of stroke, deep vein thrombosis (DVT), and/or pulmonary embolus (PE))
5. Symptomatic congestive heart failure (NYHA Class III - IV), unstable angina pectoris, cardiac arrhythmia
6. The presence of consistently abnormal laboratory values which are considered clinically significant. In addition, no subject with liver enzymes (ALT or AST) above 2 times the ULN, total bilirubin above 2 times the ULN, or serum creatinine above 1.5 ULN will be admitted to the study
7. Received an investigational drug within a period of 90 days prior to enrollment in the study
8. Received the study medication previously
9. Currently taking testosterone, testosterone-like agents, or antiandrogens,including 5-alpha reductase inhibitors (may be eligible if allow a 6 week washout period after stopping antiandrogens);
10. History of prior treatment of cancer chemotherapy agent (other than hormone therapy) or radiopharmaceutical for prostate cancer.
11. Have taken ketoconazole within the previous 12 months prior to randomization into this study
12. Have taken diethylstilbestrol or other estrogen products, ketoconazole, or abiraterone within the previous 12 months prior to randomization into this study
13. Have taken body building or fertility supplements within 4 weeks of admission into the study
14. Have been previously diagnosed with cancer (other than prostate cancer, superficial bladder cancer, or non-melanoma skin cancer).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Steiner, MD, Study Director — GTx
Locations (7):
- United States (7):
  - GTx Investigative Site, San Bernardino, California
  - GTx Investigational Site, Jeffersonville, Indiana
  - GTx Investigative Site, Albuquerque, New Mexico
  - GTx Investigative Site, Syracuse, New York
  - GTx Investigative Site, Bala-Cynwyd, Pennsylvania
  - GTx Investigative Site, San Antonio, Texas
  - GTx Investigative Site, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 subjects were enrolled with 7 subjects screen failing and 2 subjects randomized but not treated, for a total of 11 subjects treated. Outputs generated from previous company only provided data for the 11 subjects randomized. Program was halted.
Period: Overall Study
Arm/Group | 1000 mg GTx-758 BID
Started | 18
Randomized | 11
Treated | 9
Completed | 0
Not Completed | 18
Not completed — Adverse Event | 2
Not completed — Study terminated by Sponsor | 7
Not completed — Screen failure | 7
Not completed — Randomized not Treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | 1000 mg GTx-758 BID
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (10.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Decline in Serum PSA
Time Frame: 30 days
Population: Treated Patients
Measure: Count of Participants; unit: Participants
Arm/Group | 1000 mg GTx-758 BID
Number analyzed (Participants) | 9
Participants
  2 consecutive 50% or more decline | 3
  1 50% or more decline without confirmation in next visit | 1
  No 50% or more decline observed | 5

ADVERSE EVENTS:
Arm/Group | 1000 mg GTx-758 BID
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1000 mg GTx-758 BID (N=9)
Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1000 mg GTx-758 BID (N=9)
Diarrhoea (Gastrointestinal disorders) | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No